CLINICAL TRIAL: NCT02479581
Title: The Safety and Efficacy of the Enhanced Recovery After Surgery(ERAS) Applied on Cardiac Surgery With Cardiopulmonary Bypass: a Single Center, Randomized, Controlled Clinical Study
Brief Title: The Safety and Efficacy of the Enhanced Recovery After Surgery(ERAS)Applied on Cardiac Surgery With Cardiopulmonary Bypass
Acronym: ERAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: liman20150516
Record Dates: First submitted 2015-06-12; First posted 2015-06-24 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-02

CONDITIONS: Valvular Heart Disease
Keywords: Enhanced Recovery after Surgery
MeSH Terms: conditions — Heart Valve Diseases | interventions — Methylprednisolone Hemisuccinate; Scopolamine; Morphine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ERAS group (Experimental): Perioperative management follows the Enhanced Recovery after Surgery（ERAS） program
  Interventions: Procedure: ERAS group
- Conventional control group (Experimental): Perioperative management follows the conventional program
  Interventions: Procedure: ERAS group; Procedure: Conventional control group

INTERVENTIONS:
Procedure: ERAS group — Intravenous infusion of flucloxacillin sodium 1g an hour before operation
  Other Names: "yifen®","Flucloxacillin"
  Arms: ERAS group
Procedure: ERAS group — 1. No routine bowel preparation;
  2. Normal eating 1 days before the operation;
  3. No drinking 2h and solid food 6h before the operation;
  4. Drink 10% glucose 250ml 3h before operation ;
  5. Gastric mucosal protective agent was given 3 days before operation(Esomeprazole Magnesium Enteric-coated tablets 40mg/d);
  Arms: ERAS group
Procedure: ERAS group — Emphasize the preoperative psychological preparation for patients.
  Arms: ERAS group
Procedure: ERAS group — Received subcutaneous recombinant human erythropoietin (rhEPO)150（international unit/kg） once very two days from 2 days after hospital admission to 5 days postoperatively；
  Other Names: Recombinant Human Erythropoietin
  Arms: ERAS group
Procedure: ERAS group — No scopolamine and morphine before surgery; No midazolam; No anti - choline drugs;
  Arms: ERAS group
Procedure: ERAS group — Solu-Medrol®:5mg/kg intravenous infusion during the surgery;
  Other Names: "Methylprednisolone"，"Solu-Medrol® "
  Arms: ERAS group
Procedure: ERAS group — 1. Apply Transesophageal Echocardiography（TEE）after anesthesia induction;
  2. Goal-directed fluid management.
  Arms: ERAS group
Procedure: ERAS group — 1. Infusion of Human Albumin Grifol®20% 50ml;
  2. Ultrafiltration(TERUMO CARDIOVASCULAR SYSTEMS (TERUMO®));
  3. Shorten the Cardio-pulmonary Bypass line；
  4. Continuous near infrared spectrum monitoring of cerebral oxygen saturation(MNIR-P100（chongqingmingxi®）)
  Other Names: Cardio-pulmonary Bypass measures, during the surgery
  Arms: ERAS group
Procedure: ERAS group — Monitor urine volume closely, over 0.5ml/kg·h.
  Other Names: Kidney protection measure during the surgery
  Arms: ERAS group
Procedure: ERAS group — Protective ventilation strategy：Low tidal volume about 6~8ml/kg and positive end expiratory pressure（PEEP） combined with lung recruitment maneuver
  Other Names: Lung protection measure during the surgery（Dräger Primus）
Procedure: ERAS group — 1. Bilateral thoracic paravertebral block before induction of anesthesia;
  2. Fast channel anesthesia:
     * Induction use Sufentanil 0.5~1ug/kg, Vecuronium for Injection 0.15mg/kg and Etomidate 0.2~0.6mg/kg; ②. Maintain use Remifentanil Hydrochloride for Injection 0.1~0.4ug/kg·min, Propofol Injection 2~6mg/kg·h, Sevoflurane 0.5~1.5（minimum alveolar concentration） and Infusing Dexmedetomidine which load dose 0.5μg/kg in 10min then changed into 0.5-1.0μg/kg·h,Vecuronium 0.06~0.12mg/kg·h; ③. Intravenous hydromorphone Hydrochloride Injection 0.15mg/kg before surgery over.
  Other Names: Anesthesia drugs during the surgery
  Arms: ERAS group
Procedure: ERAS group — 1. Drink water after 6h, 200ml once, 2~3 times / day，
  2. early ambulation，mobilization within 48 h,
  3. Intravenous the conventional antiemetic drugs Tropisetron hydrochloride Injection 12mg qd；
  4. Intravenous the lansoprazole 30mg q12h.
  Other Names: Gastrointestinal protection measures after the surgery
  Arms: ERAS group
Procedure: Conventional control group — Routine preoperative psychological preparation for patients.
  Arms: Conventional control group
Procedure: ERAS group — After operation use Ropivacaine 100mg infiltrating intercostal wound and self-controlled intravenous analgesia pump is applicable(Sufentanil 0.05ug/kg·h combine with Ketamine 40ug/kg·h).
  Other Names: Analgesia drugs after the surgery
  Arms: ERAS group
Procedure: Conventional control group — 1. Routine bowel preparation;
  2. Liquid food eating 2 days before the operation;
  Arms: Conventional control group
Procedure: Conventional control group — Intramuscular injection of scopolamine 0.3mg combined with morphine 10mg before surgery;
  Other Names: scopolamine and morphine
  Arms: Conventional control group
Procedure: Conventional control group — 1. Induction use Sufentanil 0.5~1ug/kg, Vecuronium 0.15mg/kg and Etomidate 0.2~0.6mg/kg,Midazolam0.05~0.1mg/kg ;
  2. Maintain use Sufentanil 1~2ug/kg·h, Propofol 4~12mg/kg·h, Sevoflurane 1~3(minimal alveolar concentration)， Vecuronium 0.06~0.12mg/kg·h;
  Other Names: Routine use of anesthesia medicine during the surgery
  Arms: Conventional control group
Procedure: Conventional control group — Use self-controlled intravenous analgesia pump containing Sufentanil 0.07ug/kg·h
  Other Names: Routine use of anesthesia medicine after the surgery
  Arms: Conventional control group
Procedure: Conventional control group — Intravenous infusion of dexamethasone 20mg during the surgery
  Other Names: Dexamethasone
  Arms: Conventional control group
Procedure: Conventional control group — Intravenous infusion of flucloxacillin sodium 1g before the operation
  Other Names: "yifen®","Flucloxacillin"
  Arms: Conventional control group

SUMMARY:
This study evaluates the enhanced recovery after surgery (ERAS) concept over conventional postoperative care in patients with heart valve disease undergoing cardiac surgery with cardiopulmonary bypass. Half of participants will adherence to the ERAS, while the other half will under the conventional postoperative care.

DETAILED DESCRIPTION:
Enhanced recovery after surgery (ERAS) or fast-track surgery is a perioperative and postoperative care concept initiated in the early 1990s aiming to reduce the length of hospital stays following elective abdominal surgery. The success of ERAS depends highly on multidisciplinary teamwork and patient compliance.

This study intends to compare the Enhanced Recovery After Surgery (ERAS) concept applied to patients with heart valve disease undergoing cardiac surgery with cardiopulmonary bypass under traditional perioperative management of patients, committed to reducing patient's physical and psychological stress by surgical trauma, achieve the purpose of fast recovery, in order to establish an effective perioperative management during cardiopulmonary bypass surgery, improve patients' satisfaction and to accelerate postoperative rehabilitation safely.

ELIGIBILITY:
Inclusion Criteria:

* Heart function grade II - III (Using the cardiac function classification method formulated by American Heart Disease Institute)
* The in - hospital was treated with extracorporeal circulation operation and general anesthesia.
* Had a good cognition, and signed the informed consent.
* Aged between 18 and 70.
* The age, clinical examination and other generally situation of the two groups of patients had no statistical significance.

Exclusion Criteria:

* Combined with other blood coagulation dysfunction, serious brain, liver and kidney dysfunction, endocrine system diseases and serious infectious disease.
* Patients with severe mental disorders cannot cooperate with the treatment.
* Emergency operation
* Have taboo of Echocardiography and pulmonary catheterization by echocardiography.
* Patients have been fitted with a pacemaker.
* Allergic to erythropoietin.
* Suspected or had alcohol, drug abuse history.
* Spinal deformity or paravertebral lesions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The postoperative hospital time | From pre-surgery to discharge, up to 4 weeks
Length of ICU stay | From entering the ICU to roll out, up to 4 weeks
The time of readiness to discharge | From pre-surgery to discharge, up to 4 weeks
The length of hospital stay | From pre-surgery to discharge, up to 8 weeks
Hospitalization cost | When the patient is discharged

SECONDARY OUTCOMES:
Perioperative major adverse events | From pre-surgery to discharge, up to 4 weeks
Vasoactive drugs Support Hours | From the start of drugs to stop them, up to 4 weeks
Postoperative tracheal tube time | From the end of surgery to the removal of tracheal tube, up to 4 weeks
Duration of mechanical ventilation after surgery | From the end of surgery to the recovery of spontaneous breathing, up to 4 weeks
Time to first bowel movement | From the end of surgery to first exhaust, up to 2 weeks
Postoperative time to first exhaust | From the end of surgery to first exhaust, up to 2 weeks
Hemoglobin | baseline and 5 days after operation
  1day before and 1-5days after operation
C-reactive protein | baseline and 5 days after operation
  1day before and 1-5days after operation
Procalcitonin | baseline and 5 days after operation
  1day before and 1-5days after operation
N-terminal B-type natriuretic peptide（NT-proBNP) | baseline and 5 days after operation
  1day before and 1-5days after operation
Serum Creatinine | baseline and 5 days after operation
  1day before and 1-5days after operation
Troponin I | baseline and 5 days after operation
  1day before and 1-5days after operation
Erythrocyte Sedimentation Rate | baseline and 5 days after operation
  1day before and 1-5days after operation

OTHER OUTCOMES:
Questions to the participants' health | Six month

CONTACTS AND LOCATIONS:
Overall Officials: e wang, phD, Study Director — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

REFERENCES:
- [Result] Bakker N, Cakir H, Doodeman HJ, Houdijk AP. Eight years of experience with Enhanced Recovery After Surgery in patients with colon cancer: Impact of measures to improve adherence. Surgery. 2015 Jun;157(6):1130-6. doi: 10.1016/j.surg.2015.01.016. Epub 2015 Mar 16. PMID 25791027
- [Result] Hoffmann H, Kettelhack C. Fast-track surgery--conditions and challenges in postsurgical treatment: a review of elements of translational research in enhanced recovery after surgery. Eur Surg Res. 2012;49(1):24-34. doi: 10.1159/000339859. Epub 2012 Jul 11. PMID 22797672
- [Result] Kehlet H, Dahl JB. Anaesthesia, surgery, and challenges in postoperative recovery. Lancet. 2003 Dec 6;362(9399):1921-8. doi: 10.1016/S0140-6736(03)14966-5. PMID 14667752
- [Derived] Li M, Zhang J, Gan TJ, Qin G, Wang L, Zhu M, Zhang Z, Pan Y, Ye Z, Zhang F, Chen X, Lin G, Huang L, Luo W, Guo Q, Wang E. Enhanced recovery after surgery pathway for patients undergoing cardiac surgery: a randomized clinical trial. Eur J Cardiothorac Surg. 2018 Sep 1;54(3):491-497. doi: 10.1093/ejcts/ezy100. PMID 29514224